CLINICAL TRIAL: NCT00119626
Title: SAINT I (Stroke - Acute Ischemic - NXY Treatment) A Double Blind, Randomized, Placebo Controlled, Parallel Group, Multicenter, Phase IIb/III Study to Assess the Efficacy and Safety of Intravenous NXY-059 in Acute Ischemic Stroke.
Brief Title: Safety and Effectiveness of NXY-059 for the Treatment of Patients Who Have Suffered From a Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SA-NXY-0006; 0006; SAINT I
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Cerebral Stroke; Ischemic Attack, Transient
Keywords: Stroke, Acute; Cerebrovascular Stroke
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — disufenton sodium

INTERVENTIONS:
Drug: NXY-059

SUMMARY:
This study will determine if NXY-059 will reduce functional disability from an acute stroke. The study is designed to look at both overall recovery and recovery of motor function, for example muscle strength and coordination.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Acute ischemic stroke with limb weakness, onset of symptoms within 6 hours
* Full functional independence prior to the present stroke

Exclusion Criteria:

* Unconsciousness
* Subjects who are unlikely to complete the infusion of investigational product and/or are unlikely to undergo active medical management during that period due to a severe clinical condition
* Severe illness with life expectancy less than 6 months
* Known severe kidney disorder
* Current known alcohol or illicit drug abuse or dependence
* Pregnant or breast-feeding
* Treatment with acetazolamide and methotrexate is not permitted during the infusion
* Participation in a previous clinical study within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700
Dates: Start 2003-06; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Global disability on modified Rankin scale at 90 days.

SECONDARY OUTCOMES:
NIH stroke scale (termed "co-primary" in study protocol), Barthel Index, Stroke Impact Scale, EQ-5D all at 90 days, Safety outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca NXY-059 Medical Science Director, MD, Study Director — AstraZeneca
Locations (2):
- Research Site, Södertälje, Sweden
- Research Site, Glasgow, United Kingdom

REFERENCES:
- [Result] Lees KR, Zivin JA, Ashwood T, Davalos A, Davis SM, Diener HC, Grotta J, Lyden P, Shuaib A, Hardemark HG, Wasiewski WW; Stroke-Acute Ischemic NXY Treatment (SAINT I) Trial Investigators. NXY-059 for acute ischemic stroke. N Engl J Med. 2006 Feb 9;354(6):588-600. doi: 10.1056/NEJMoa052980. PMID 16467546